CLINICAL TRIAL: NCT05788081
Title: Treatment Of Newly-diagnosed Follicular Lymphoma With CELMoD Golcadomide, Rituximab +/- Nivolumab: An Umbrella Bayesian Optimal Phase II Study.
Brief Title: Treatment Of Newly-diagnosed Follicular Lymphoma With CELMoD Golcadomide, Rituximab +/- Nivolumab.
Acronym: TOP-FLOR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Austin Health (Other Government); Grampians Health (Unknown); Fiona Stanley Hospital (Other); Eastern Health (Other); Barwon Health (Other Government); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM048-1036
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Follicular Lymphoma Stage II; Follicular Lymphoma Stage III; Follicular Lymphoma Stage IV
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Nivolumab; Rituximab

STUDY DESIGN:
Intervention Model Description: Study Design Open label multicentre umbrella Bayesian Optimal Phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A- Golcadomide + Rituximab (Experimental): Rituximab 375mg/m2 IV infusion Q4W + golcadomide 0.4mg po D1-D14 of each cycle for 8 cycles, followed by Rituximab 375mg/m2 IV infusion Q12W in participants with CR/PR at end of induction
  Interventions: Drug: golcadomide; Drug: Rituximab
- Arm B- Nivolumab + golcadomide + Rituximab (Experimental): Nivolumab 480mg IV infusion Q4W, Rituximab 375mg/m2 IV infusion Q4W and golcadomide 0.4mg po D1-D14 of each cycle for 8 cycles, followed by Rituximab 375mg/m2 IV infusion Q12W in participants with CR/PR at end of induction
  Interventions: Drug: golcadomide; Drug: Nivolumab 10 MG/ML; Drug: Rituximab

INTERVENTIONS:
Drug: golcadomide — BMS-986369 is an orally administered Cereblon-modulating compound
  Other Names: BMS-986369; CC-99282
Drug: Nivolumab 10 MG/ML — Nivolumab is a fully humanised IgG4 blocking monoclonal antibody against PD-1.
  Other Names: Opdivo
  Arms: Arm B- Nivolumab + golcadomide + Rituximab
Drug: Rituximab — Rituximab is a chimeric anti-CD20 antibody containing human IgG lambda and kappa constant regions with murine variable regions
  Other Names: Mabthera

SUMMARY:
First line treatment with combination rituximab and golcadomide with, or without nivolumab, in patients in previously untreated Follicular Lymphoma

DETAILED DESCRIPTION:
This study will involve participants with a condition called Follicular Non Hodgkin Lymphoma (Follicular Lymphoma).

The main purpose of this study is to see if it is safe to give an induction schedule of the drug golcadomide, in combination with Rituximab +/- Nivolumab, and to see how effective this combination is in patients who have had no previous drug treatment for their lymphoma. In particular, we will be monitoring for any specific side effects which may be increased by adding golcadomide to Rituximab treatment +/- Nivolumab for 8 cycles (28 days per cycle), with up to 2 years of maintenance treatment of rituximab in eligible patients following induction.

Participants will be reviewed at baseline and prior to each cycle of treatment for toxicity, scans will be performed at baseline, after 2 and 5 cycles of induction treatment, and every 8 weeks during maintenance phase. Following completion of treatment, participants will be followed up for a total of 3 years (every 6 months). In participants with relapsed disease, these will be followed for survival every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+ years.
2. Histologically proven CD20 positive Follicular non Hodgkin lymphoma (FL) grades 1-3A (i.e. classical follicular lymphoma according to the current World Health Organization classification).3
3. No previous chemotherapy, or other investigational drug for this indication apart from focal radiotherapy.
4. Stage II-IV disease (Ann Arbor criteria).
5. Eastern Collaborative Oncology Group (ECOG) performance status 0 to 1 unless attributable to lymphoma, in which case patients of performance status 2 are also eligible.
6. Measurable FDG avid disease on baseline PET/CT scan.
7. Deemed to need treatment by treating investigator. Reasons for treatment can include, but are not limited to:

a. Any nodal or extranodal tumour mass >7cm AND/OR multiple extranodal disease sites b. Involvement of at least 3 sites each with diameter >3cm c. Symptomatic splenic enlargement d. Organ involvement/compression e. Ascites or pleural effusion f. Lactate Dehydrogenase (LDH) elevated g. Presence of systemic symptoms h. Disease progression in preceding 3 months i. Evidence of marrow infiltration with marrow compromise. (e.g., Hb, WCC or plt count below lower limit of institutional normal range).

h) Adequate bone marrow function including:

1. Haemoglobin >8.0 g/dL
2. White cell count (WCC) ≥2000/μL
3. Neutrophils >1.5 x 109/L
4. Platelets >75 x 109/L at the time of study entry, unless attributed to bone marrow infiltration by lymphoma.

i) Adequate renal function with serum creatinine ≤1.5 x ULN or creatinine clearance (CrCl) ≥ 60mL/min (using Cockcroft-Gault formula, 24hr urine collection or eGFR).

Female CrCl = (140 - age in years) x weight (kg) x 0.85 72 x serum creatinine (mg/dL)

Male CrCl = (140 - age in years) x weight (kg) x 1.00 72 x serum creatinine (mg/dL) j) Adequate hepatic function with AST/ALT ≤3x ULN and total bilirubin ≤1.5 x ULN (except subjects with Gilbert syndrome, who can have a total bilirubin ≤3 mg/dL or ≤51.3 μmol/L).

k) Adequate left ventricular ejection fraction of >45% as demonstrated on a Gated Cardiac Blood Pool Scan or echocardiogram.

l) Life expectancy > 3 months. m) Patients of childbearing potential willing to adhere to the following contraceptive precautions.

1. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
2. Females must not be breastfeeding.
3. FCBP must use appropriate method(s) of contraception to avoid pregnancy for 23 weeks (30 days plus five half-lives of nivolumab) and 28 days for golcadomide post-treatment completion.
4. Men who are sexually active with FCBP must use any contraceptive method with a failure rate of less than 1% per year. They must agree to adhere to contraception for a period of 90 days from the last day golcadomide and refrain from donating sperm.
5. Azoospermic males and FCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.

m) Written, informed consent.

Exclusion Criteria:

1. Follicular large B-cell Lymphoma (Grade 3B) transformed follicular lymphoma, other indolent lymphomas.
2. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
3. Central nervous system, meningeal involvement or spinal cord compression by lymphoma.
4. Patients with active, known or suspected autoimmune disease. Patients with well controlled type I diabetes mellitus, coeliac disease, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, vitiligo or psoriasis not requiring systemic treatment, or other conditions not expected to recur in the absence of an external trigger are permitted to enrol.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement therapy are permitted in the absence of active autoimmune disease.
6. Past history of interstitial lung disease.
7. Prior organ transplantation or allogeneic bone marrow transplantation.
8. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
9. Uncontrolled or severe cardiovascular disease (NYHA class III or IV heart failure; myocardial infarction within the last 6 months of study entry); unstable angina; unstable cardiac arrhythmias; clinically significant pericardial disease.
10. Any other serious active disease.
11. Any positive test result for hepatitis B or hepatitis C virus during screening indicating acute or chronic infection. Latent hepatitis B with undetectable viral load by PCR is allowable provided appropriate anti-viral prophylaxis is given as per institutional guidelines.
12. Any positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
13. Any history of severe hypersensitivity reactions to other monoclonal antibodies.
14. A history of allergy or intolerance (unacceptable AEs) to study drug components or Polysorbate-80-containing infusions.
15. Medical or psychiatric conditions that compromise the patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve a complete metabolic response in the absence of prohibitive toxicity with induction rituximab, golcadomide with or without nivolumab comprising 8 cycles of therapy with each cycle delivered every 4 weeks. | Consent to 8 weeks after last induction treatment (maximum 44 weeks)
  Metabolic response as assessed by PET/CT and defined by Lugano criteria; toxicities as defined by CTCAE v5

SECONDARY OUTCOMES:
To assess overall toxicity | Day 1 to 30 days after the end of maintenance phase (up to maximum 32 months)
  As determined by rate of toxicity grade 3 or higher per CTCAE V5
To assess time to treatment failure | Day 1 end of follow up period (up to a maximum of 5 years)
  Treatment response assessed by PET/CT according to the Lugano classification for Response Criteria for Non-Hodgkin Lymphoma
Progression free survival | Day 1 end of follow up period (up to a maximum of 5 years)
  Quantification of progression free survival
Overall survival | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  Quantification of OS

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Hawkes, MBBS, Principal Investigator — Austin Health
Locations (5):
- Australia (5):
  - Grampians Health, Ballarat, Victoria
  - Eastern Health, Box Hill, Victoria
  - University Hospital Geelong, Barwon Health, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No